CLINICAL TRIAL: NCT00099541
Title: A Dual-Cohort, Prospective, Observational Study of Unresectable Stage IIIB/IV Non-Small Cell Lung Cancer Patients With and Without Bone Metastasis
Brief Title: Non-small Cell Lung Cancer Registry
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EUS99; US99; Z-NEXT
Record Dates: First submitted 2004-12-15; First posted 2004-12-16 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Non-Small-Cell Lung Cancer; Pleural Effusion, Malignant
Keywords: Lung Cancer; Bone Metastases; Bone Markers; NTX; zoledronic acid; Registry; Unresectable Stage IV Non Small-cell Lung Cancer (NSCLC); Unresectable Stage IIIB NSCLC with Pleural Effusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant; Lung Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
This trial will evaluate two separate groups of patients with stage IIIB/IV non-small cell lung cancer. The objective of Group 1 is to investigate an FDA-approved drug in stage IIIB/IV non-small cell lung cancer patients that has spread to the bones. The objective of Group 2 is to see if a blood test can be used to predict when cancer-related bone lesions develop. This trial is seeking patients 18 years or older that have been diagnosed with Stage IIIB or Stage IV non-small cell lung cancer that cannot be treated by surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Histologically confirmed NSCLC (squamous cell carcinoma, adenocarcinoma, large cell carcinoma).
* Unresectable Stage IIIB with pleural effusion or stage IV NSCLC
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Patients who received an IV bisphosphonate (e.g.pamidronate; zoledronic acid)
* Patients who received an oral bisphosphonate therapy in the 6 months prior to screening (alendronate; etidronate; risedronate; tiludronate; ibandronate)
* Patients who are currently receiving any investigational drugs that are suspected to have renal toxicity and/or are excreted by the kidneys
* Known clinically significant hypersensitivity to zoledronic acid or other bisphosphonates or any of the excipients in the formulation of zoledronic acid (mannitol, sodium citrate)
* Abnormal renal function or creatinine clearance
* Unstable brain metastasis
* Women of childbearing potential not using a medically recognized form of contraception, as well as women who are breastfeeding
* Patients with nonmalignant conditions which would confound the evaluation of the primary endpoint, impair tolerance of therapy, or prevent compliance to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-11; Study Completion 2007-11

PRIMARY OUTCOMES:
Group 1: Time to the first occurrence of an skeletal related event (SRE) in unresectable stage IIIB/IV NSCLC patients with bone metastases
Group 2: Observational

SECONDARY OUTCOMES:
Patients with an SRE will be evaluated for:
Time from stage IIIB/IV NSCLC diagnosis to progression to bone
Time from bone metastasis diagnosis to presentation of clinical symptoms of skeletal complications
The effect of serum NTX levels on the development of skeletal events (SREs), and
Overall survival
Group 2: Obervational

CONTACTS AND LOCATIONS:
Overall Officials: L. Lacerna, MD, Study Chair — Novartis Pharmaceuticals
Locations (101):
- United States (101):
  - Birmingham Hematology and Oncology Associates, Birmingham, Alabama
  - Hembree Cancer Center-St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Pacific Cancer Medical Center Inc., Anaheim, California
  - Bay Area Cancer Research Group, Concord, California
  - Fresno Hem/Onc Medical Group, Fresno, California
  - Beaver Med Group, Highland, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - Stockton Hem. Onc., Stockton, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Greeley Medical Clinic, Greeley, Colorado
  - Western Hematology/Oncology, Lakewood, Colorado
  - Hematology Oncology PC, Stamford, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Gainesville Hematology Oncology Associates, Gainesville, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - Center for Cancer Care & Research, Lakeland, Florida
  - Lake Heart & Cancer Center, Leesburg, Florida
  - Melbourne Internal Medicine Assoc (MIMA) Century Research, Melbourne, Florida
  - Pasco Pinellas Cancer Center, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Mid- Florida Hematology & Oncology Centers, PA, Orange City, Florida
  - Space Coast Medical, Titusville, Florida
  - Vero Beach Hematology/Oncology, Vero Beach, Florida
  - Hematology & Oncology of N.E. GA, Athens, Georgia
  - Augusta Onc. Associates, Augusta, Georgia
  - Suburban Hematology-Oncology, Snellville, Georgia
  - Regional Cancer Center, Danville, Illinois
  - The Cancer Institute at Alexian Brothers, Elk Grove Village, Illinois
  - Lekha Babu M.D Ltd., Flossmoor, Illinois
  - Joliet Oncology Hematology Associates, Ltd, Joliet, Illinois
  - LaGrange Oncology Associates, LaGrange, Illinois
  - Northwest Medical Specialists, Niles, Illinois
  - Midwest Cancer Research Group, Skokie, Illinois
  - Medical Consultants, PC, Muncie, Indiana
  - Kentuckiana Cancer Center, PLLC, Louisville, Kentucky
  - W. Kentucky Hematology's Oncology Group, PSC, Paducah, Kentucky
  - Cabrini Center for Cancer Care, Alexandria, Louisiana
  - Louisiana Oncology Associates, Lafayette, Louisiana
  - Hematology and Oncology Specialists, Metairie, Louisiana
  - Highland Clinic, APMC, Shreveport, Louisiana
  - Sinai Hospital, Baltimore, Maryland
  - Maryland Hematology/Oncology Associates, Baltimore, Maryland
  - David H. Smith, MD, Chestertown, Maryland
  - Oncology-Hematology Associates, PA, Clinton, Maryland
  - Maryland Oncology, Columbia, Maryland
  - St. Joseph Medical Center, Towson, Maryland
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - Fallon Clinic, Worcester, Massachusetts
  - Henry Ford Medical Center, Detroit, Michigan
  - Singh & Arora Hematology/Oncology, Flint, Michigan
  - Hubert Humphrey Cancer Center, Robbinsdale, Minnesota
  - Heartland Hematology/Oncology Associates Inc., Kansas City, Missouri
  - St. Joseph Onocology, Inc., Saint Joseph, Missouri
  - University Hematology Oncology, Inc., St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Sierra Nevada Oncology Care, Carson City, Nevada
  - Nevada Cancer Center, Las Vegas, Nevada
  - US Oncology, Las Vegas, Nevada
  - Center For Cancer & Hematologic Disease, Cherry Hill, New Jersey
  - HOANNJ/Carol G. Simon Cancer Center, Morristown, New Jersey
  - Medical Hematology/Oncology, Somerset, New Jersey
  - Hematology-Oncology Associates of CNY, East Syracuse, New York
  - Huntington Medical Group, Huntington Station, New York
  - Broome Oncology, Johnson City, New York
  - Kin Yui Lam, MD, New York, New York
  - Alamance Regional Medical Ctr. Cancer Ctr., Burlington, North Carolina
  - Raleigh Hematology Oncology Associates, Raleigh, North Carolina
  - Summa Health System, Akron, Ohio
  - OHCI, Cincinnati, Ohio
  - Mukesh Bhatt, MD, Medina, Ohio
  - Lawrence M. Stallings, MD, LLC, Wooster, Ohio
  - M. Farouk Kanaa, MD, Inc., Oklahoma City, Oklahoma
  - Cancer Treatment Center, Tulsa, Oklahoma
  - Oncology-Hematology of Lehigh Valley PC, Bethlehem, Pennsylvania
  - Paul V. Woolley MD PC, Johnstown, Pennsylvania
  - Chester County Hematology/Oncology Services, West Chester, Pennsylvania
  - South Carolina Oncology Assoc., PA, Columbia, South Carolina
  - Palmetto Hematology Oncology, P.C, Spartanburg, South Carolina
  - Associates in Oncology and Hematology, Chattanooga, Tennessee
  - The Family Cancer Center, PLLC, Collierville, Tennessee
  - McLeod Cancer & Blood Center, Johnson City, Tennessee
  - Kingsport Hematology-Oncology, Kingsport, Tennessee
  - Eastern Connecticut Hematology/Oncology, Memphis, Tennessee
  - Oncology Hematology of South Florida, Memphis, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Southwest Regional Cancer Center, Austin, Texas
  - St. Joseph Regional Cancer Ctr., Bryan, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Center for Oncology Research and Treatment, PA, Dallas, Texas
  - Oncology Consultants P.A., Houston, Texas
  - South Texas Oncology & Hematology, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Cancer Outreach, Abingdon, Virginia
  - Lynchburg Oncology, Lynchburg, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Oncology/Hematology Association of SW VA, Roanoke, Virginia
  - Western WA Med. Grp. Oncology, Everett, Washington
  - Western Washington Oncology, Lacey, Washington
  - Swedish Health Services, Seattle, Washington
  - Oncology Alliance, S.C., Glendale, Wisconsin

REFERENCES:
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com